CLINICAL TRIAL: NCT02993016
Title: Comparison of Conventional Versus Patient-specific Instruments in Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Conventional Versus Patient-specific Instruments in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: patient-specific instruments
Record Dates: First submitted 2016-12-08; First posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Osteoarthritis, Patient-specific Instruments
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- patient-specific instruments group (Experimental): procedure: PSI (patient-specific instruments) will be used as the cutting guide in total knee arthroplasty.
  Interventions: Procedure: patient-specific instruments; Device: The Signature™ Vanguard
- conventional instruments group (Active Comparator): procedure: Conventional instruments will be used as the cutting guide in total knee arthroplasty.
  Interventions: Procedure: conventional instruments; Device: Vanguard PS(posterior stabilized)

INTERVENTIONS:
Procedure: patient-specific instruments
  Arms: patient-specific instruments group
Device: The Signature™ Vanguard
  Arms: patient-specific instruments group
Procedure: conventional instruments
  Arms: conventional instruments group
Device: Vanguard PS(posterior stabilized)
  Arms: conventional instruments group

SUMMARY:
Total knee arthroplasty (TKA) has a high success rate for addressing pain and improving function. However, in instances where incorrect positioning and malignment of the TKA components are observed, patients can experience a range of negative postoperative outcomes such as loss of thickness of polyethylene tibial bearings, eccentric loading, implant loosening, and eventual early revision. To avoid these complications, achieving a postoperative alignment within the range of 0°±3° of the mechanical axis is recommended. Manual intramedullary/extramedullary guides are not thought to be capable of consistently achieving axes in this range, and though computer-assisted navigation has shown superior results in comparison with conventional instrumentation, it is also limited by increased surgical times and no clear superiority in improving short-term clinical outcomes. Thus, there has been in a push in the orthopaedic community to create more precise technologies to aid in the reconstruction of the knee's mechanical axis. Patient-specific instrumentation (PSI), which uses anatomical data obtained primarily from pre-operative axial computed tomography (CT) or magnetic resonance imaging (MRI) to create disposable cutting jigs individualized to the patient's unique anatomy, was created with this goal.

This study aims to compare the clinical results of conventional and patient-specific instruments in total knee arthroplasty.

DETAILED DESCRIPTION:
The objective of this work was to compare pain, stiffness, function and accuracy between groups at minimum 2 year postoperatively. The investigators hypothesized that PSI would lead to a neutral mechanical axis on average more frequently than conventional instrumentation.

The study design is a double-blind randomized controlled trial. Randomly, fifty patients planed to undergo total knee arthroplasty using conventional instruments and other fifty patients undergo total knee arthroplasty using patient-specific instruments. The clinical outcome is comparative preoperative, postoperative 6weeks, 3months, 6months and 1years. And clinical score consists of Range of Motion (ROM), WOMAC (Western Ontario and McMaster University Arthritis Index) pain scale (preoperative and postoperative 6, 12, 24 months), Knee Society Score (preoperative and postoperative 6, 12, 24 months), Anterior and posterior stress view on X-ray (preoperative and postoperative 6, 12, 24 months).

ELIGIBILITY:
Inclusion Criteria:

* over 19 year old
* Patients for total knee arthroplasty of both knee
* over 5 degree in lateral bowing of femur
* having medicare insurance

Exclusion Criteria:

* Rheumatoid arthritis
* Other inflammatory arthritis
* Neuropsychiatric patients
* Hepatic insufficiency
* Renal insufficiency
* over 40 of body mass index
* Chronic opioid use (taking opioids for longer than 3 months)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Range of Motion (ROM) | Changes from Baseline Range of Motion at postoperative 1 year

SECONDARY OUTCOMES:
Changes in WOMAC (Western Ontario and McMaster University Arthritis Index) | Changes from Baseline score to score of postoperative 1 year
Changes in Knee Society Score | Changes from Baseline score to score of postoperative 1 year
Changes in Anterior and posterior stress view on X-ray | Changes from Baseline Anterior and posterior stress view on X-ray at postoperative 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yong In, MD, PhD, Study Chair — the Catholic Univerisity of Korea Seoul St Mary's hospital

REFERENCES:
- [Derived] ALShammari SA, Choi KY, Koh IJ, Kim MS, In Y. Total knee arthroplasty in femoral bowing: does patient specific instrumentation have something to add? A randomized controlled trial. BMC Musculoskelet Disord. 2021 Apr 2;22(1):321. doi: 10.1186/s12891-021-04198-5. PMID 33794854